CLINICAL TRIAL: NCT04911465
Title: Continuous Assessment of Hemodynamic Compensation in Pediatric Trauma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20-2755
Record Dates: First submitted 2021-05-24; First posted 2021-06-03 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Trauma
Keywords: Pediatric
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Pediatric Trauma Patients: All pediatric patients >31 days who meet criteria for highest level trauma activation (Level Red or Level 1) at the Children's Hospital Colorado.
  Interventions: Device: Flashback CRI T1 Tablet

INTERVENTIONS:
Device: Flashback CRI T1 Tablet — Collect continuous data on the compensatory reserve index, a measurement of a patient's central volume status.

SUMMARY:
This is an observation study using the Flashback CRI T1 tablet to collect data on compensatory reserve index in pediatric trauma patients. Highest trauma activations at the institution will be enrolled in the study and data will be collected for 12-24 hours based on the patient's hemodynamic status. The device collects data via a pulse oximeter probe. No treatment decisions will be made based on the values of the on the CRI tablet. Data will be retrospectively reviewed to determine if any trends exist that correlate with blood loss, need for operation or blood transfusion.

ELIGIBILITY:
Inclusion Criteria:

• Children 31 days through 26 years (inclusive) of age who undergo Trauma Red (highest level) activation or Trauma Level 1 (mid-level) activation at Children's Hospital Colorado or Children's National Medical Center.

Exclusion Criteria:

* Pregnant patients
* Incarcerated patients
* Patients who object to study participation at any time
* Limited access to or compromised monitoring sites for non-invasive finger sensors
* Brain death (GCS 3 with fixed, dilated pupils)

Ages: 31 Days to 26 Years | Sex: All
Age Groups: Child, Adult
Study Population: Traumatically injured pediatric patients who present to Children's Hospital Colorado or Children's National Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with abnormal CRI values | 12-24 hours
  Compare CRI values collected by the T1 tablet to standard traditional vital signs, i.e. heart rate and blood pressure, to identify if abnormal CRI values correlated with abnormal traditional vital signs
Number of participants who require blood products | 12-24 hours
  Compare CRI values collected by the T1 tablet to standard laboratory measures, i.e. hematocrit, to identify if abnormal CRI values correlated with blood loss
Number of participants who require operation or angiographic intervention | 12-24 hours
  Determine if CRI values collected by the T1 tablet are abnormal in the setting of patients who require operation or angiographic intervention for hemorrhage control

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Moulton, MD, Principal Investigator — Children's Hospital Colorado
Locations (2):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No